CLINICAL TRIAL: NCT07393100
Title: The Acute Effect of Shoulder Kinesiology Taping Application on Dental Students in the Clinic
Brief Title: The Acute Effect of Shoulder Kinesiology Taping on Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Serap Akyol, Physiotherapist, European University of Lefke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK054.02
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dominant shoulder kinesiology taping (Experimental): This study investigates the acute effects of shoulder kinesiology taping (KB) in a clinical setting among final-year dental students experiencing musculoskeletal discomfort related to their professional activities.
  Intervention:
  Participants received kinesiology taping applied to the dominant shoulder region targeting the deltoid and supraspinatus muscles. The taping was designed to provide muscular facilitation, enhance joint stabilization, and modulate pain through biomechanical and neurophysiological mechanisms. The application followed standardized protocols based on rehabilitation principles for shoulder injuries, with specific techniques including:
  Y-strip application for deltoid inhibition (to reduce overuse-related tension and pain modulation).
  I-strip applications for supraspinatus facilitation and humeral head centralization.
  Additional I-strip for acromioclavicular joint stabilization and fascial correction.
  The taping was applied in three sessions, spaced one day apar
  Interventions: Other: Kinesiology Taping

INTERVENTIONS:
Other: Kinesiology Taping — The kinesiology taping (KT) protocol applied within the scope of the study was carried out over three sessions, every other day, in accordance with the biomechanical requirements of the shoulder complex. This four-stage protocol applied to the participants lasted a total of three sessions for each participant. Throughout the application, participants were asked to continue their normal daily life activities, and final measurements were taken one day after the last session.

SUMMARY:
Research Objective and Participants' Role:

We invite you to participate in a scientific study aimed at reducing the load on your shoulder region during dental clinical practice. The main goal of this study is to scientifically examine the immediate (acute) effects of kinesiology taping applied to the shoulder region on your pain level, shoulder function, general quality of life, and job satisfaction. You have been included in this research because you are a final-year student and actively work in a clinical setting.

How Will the Application Process Proceed?

If you agree to participate, the process will consist of the following steps:

Evaluation: First, we will administer a short form regarding your age, height, weight, and clinical work pace, along with scientific questionnaires assessing your pain intensity, shoulder functionality, quality of life, and job satisfaction.

Taping: To support the deltoid and supraspinatus muscles in your shoulder region, kinesiology taping will be applied under the supervision of a physiotherapist every other day, for a total of three sessions. These tapes are skin-friendly, elastic, and designed not to restrict your movement.

Final Test: One day after the completion of the third session, you will be asked to fill out the same questionnaires again to measure the changes brought about by the taping.

Your Rights and Privacy

Voluntary Participation: Participation in this study is entirely voluntary. Even if you sign the form, you may withdraw from the study at any time without providing any reason and without facing any penalties that would affect your academic progress.

Risks and Costs: Kinesiology taping is generally a safe method, and there will be no financial cost to you for participating. No payment will be made for your participation. In the rare case of skin sensitivity during the application, please inform the researcher.

Confidentiality: Your identity will be kept completely confidential and will only be known to the researcher. The data obtained will be used in scientific publications in aggregated form, without disclosing your name.

Consent Declaration If you have read and understood this information and your questions have been answered, you may sign the form to indicate your voluntary consent to participate in the study.

DETAILED DESCRIPTION:
Research Objective and Participant Role You are invited to participate in this research because you are a final-year student at the Faculty of Dentistry, Lefke European University, and actively engaged in clinical practice. The main objective of this study is to scientifically examine the acute (short-term) effects of kinesiological taping applied to the shoulder area during clinical practice in dental students.

To this end, you will be asked to provide the following contributions:

Complete the scientific scales and questionnaires,

Agree to undergo kinesiological taping for a total of three sessions, applied every other day,

Complete the same scales again after the application.

This research aims to contribute to the development of low-cost and practical interventions to support the professional musculoskeletal health of dental students.

Research Process and Implementation Stages

If you confirm your participation, the process will consist of the following stages:

1. Preliminary Assessment (Pre-Taping):

   First, you will complete a form containing your demographic information such as your age, height, weight, clinical study duration, exercise, and smoking habits.

   Then, four different scientific scales will be administered:
   1. Visual Analog Scale (VAS): To assess the severity of your predominant shoulder pain experienced during clinical practice.
   2. Arm-Shoulder-Hand Disorders Rapid Questionnaire (QuickDASH): To measure the functionality of your upper extremity (arm, shoulder, hand) in daily activities.
   3. World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF): To assess the physical, psychological, social, and environmental dimensions of your overall quality of life.
   4. Minnesota Job Satisfaction Scale (Short Form): To determine your job satisfaction with your clinical practice.
2. Kinesiological Taping Application (Intervention):

   Kinesiological taping will be applied to support your shoulder muscles (especially the deltoid and supraspinatus) that have been overloaded during clinical practice.

   The application was performed by a physical therapist (Serap AKYOL).

   The tapes are skin-friendly, water-resistant, hypoallergenic, and elastic. They do not restrict your normal joint movement and do not interfere with your daily activities (bathing, sleeping, etc.).

   The application will be done every other day for a total of 3 sessions (e.g., Monday, Wednesday, Friday). Each session will last approximately 15-20 minutes.

   The tapes will be removed after the third session, or they may fall off on their own.
3. Final Assessment (After Taping):

The day following the third taping session, the same four scientific scales (VAS, QuickDASH, WHOQOL-BREF, Minnesota) applied in stage 1 will be reapplied.

This will be done to measure the effects of kinesiological taping on pain, function, quality of life, and job satisfaction.

Total Participation Duration: The entire process (preliminary assessment, 3 application sessions, final assessment) will take approximately 1 week.

Your Rights and Privacy

1. Voluntariness and Right to Withdraw:

   Your participation in this research is entirely voluntary.

   Even if you have signed this form, you can withdraw from the research at any time without giving any reason.

   Your withdrawal will not affect your academic status, grades, or relationship with the university in any way.
2. Risks and Costs:

   Kinesiological taping is generally a safe, non-invasive (non-surgical) method.

   You will not incur any financial burden for your participation (it is free).

   No payment will be made for your participation.

   In the very rare cases of skin irritation, redness, or itching, please report it immediately to the researcher. In such a case, the tapes will be removed and necessary recommendations will be made.
3. Privacy and Data Use:

All information regarding your identity (name, surname, student number) will be kept completely confidential and will only be known by the researchers of this study.

The collected data will be stored in a computer environment under an encrypted and anonymous (nameless) code number.

The results obtained will be used collectively and statistically in scientific publications, thesis studies, or academic presentations; your personal identification information will absolutely not be disclosed.

ELIGIBILITY:
Participant inclusion criteria:

* Being a fifth-year student at the Lefke European University Faculty of Dentistry.
* Being between 22 and 26 years of age.

Exclusion criteria for participants:

* History of acute trauma or major surgery.
* History of allergic reaction to kinesiology tape.
* Severe structural damage to the shoulder joint (dislocation, fracture, etc.).

Ages: 22 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | The study ended one week after registration. Since the application was administered three times every other day, each participant was recorded on Mondays, Wednesdays, and Fridays. The total study duration was four weeks.
  It was used to measure pain in the dominant shoulder of participants. There is a 10 cm line between two extremes: "no pain" and "extreme pain," and participants are asked to mark the intensity of their pain on this line. 0 indicates no pain, while 10 indicates unbearable pain.
Disabilities of the Arm, Sholder and Hand (Quick-DASH) | The study ended one week after registration. Since the application was administered three times every other day, each participant was recorded on Mondays, Wednesdays, and Fridays. The total study duration was four weeks.
  It was used to assess participants' upper extremity functionality in detail. Participants completed the scale subjectively. The Arm, Shoulder, and Hand Quick Survey consists of 11 items that examine the patient's health status over the past week, the degree of difficulty experienced during physical activities involving the upper extremities, the severity of symptoms such as tingling and pain, and the impact of these symptoms on social activities, sleep, or work. Scoring is done on a scale from 0 (no disability) to 100 (most severe disability), with higher scores reflecting greater disability.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) scale | The study ended one week after registration. Since the application was administered three times every other day, each participant was recorded on Mondays, Wednesdays, and Fridays. The total study duration was four weeks.
  It was used to assess participants' quality of life in detail before and after kinesiology taping. Participants completed the scale subjectively. The scale consists of 24 items covering four main areas: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items), plus two additional items assessing health satisfaction and overall quality of life. Items are scored using a 5-point Likert scale, with higher scores indicating higher quality of life. Scores range from 0-100.
Minnesota Job Satisfaction Scale | The study ended one week after registration. Since the application was administered three times every other day, each participant was recorded on Mondays, Wednesdays, and Fridays. The total study duration was four weeks.
  It was used to assess job satisfaction before and after kinesiology taping was applied to participants. Participants filled out the scale subjectively. The scale consists of 20 items and is typically rated on a 5-point Likert scale, with a high score indicating good job satisfaction. Scores range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Akyol, Principal Investigator
Locations (1):
- European University of Lefke, Lefka, Cyprus

REFERENCES:
- See also: Aboalshamat, K. T. (2020). Nordic assessment of occupational disorders among dental students and dentists in Saudi Arabia. Journal of International Society of Preventive & Community Dentistry, 10(5), 561-568. — https://pubmed.ncbi.nlm.nih.gov/33282764/
- See also: Alkadi, L. T., Masuadi, E., Mohamed, T. A., Mohamud, M. S., & Farook, F. F. (2022). A Likert scale versus a visual analogue scale and the participant response: A cross sectional study. Journal of International Dental and Medical Research, 15(1), 255-262. — https://api.semanticscholar.org/CorpusID:249878649
- See also: Almeida, M. B., Póvoa, R., Tavares, D., Alves, P. M., & Oliveira, R. (2023). Prevalence of musculoskeletal disorders among dental students: A systematic review and meta-analysis. Heliyon, 9(9), e19956. — https://pubmed.ncbi.nlm.nih.gov/37780768/
- See also: AlSahiem, J., Alghamdi, S., AlQahtani, R., AlOtaibi, N., AlMazyad, A., AlHarbi, M., AlRasheed, M., & AlAnazi, F. (2023). Musculoskeletal disorders among dental students: A survey from Saudi Arabia. BMC Oral Health, 23(1), 795. — https://jicrcr.com/index.php/jicrcr/article/view/910
- See also: Alshahrani, A. M. A., Alshehri, W. A. A., Hamdan, A. E. B., Aloufi, S. A., Almutairi, N. M. T., Hakami, A. A., Al Ali, R. A., & Alhawiti, A. A. K. (2024). Evaluation of dentists' job satisfaction through a systematic review. — https://jicrcr.com/index.php/jicrcr/article/view/910
- See also: Altaş, N., Çukurova Yılmaz, Z., & Uzun, E. V. (2022). Evaluation of the working posture and upper extremity musculoskeletal complaints among dentistry students. Turkish Journal of Public Health, 20(1), 70-79. — https://dergipark.org.tr/tr/download/article-file/1779695
- See also: Aydın, F., Özalp, B. T., & Gündüz, T. (2022). Ergonomik risk analizi yöntemleri ve metabolik hız hesabı yazılım uygulaması [Methods of ergonomic risk analysis and metabolic rate calculation software application]. Uludağ Üniversitesi Mühendislik Fakültesi — https://dergipark.org.tr/tr/download/article-file/1779695
- See also: Baltacı, G. (2015). Omuz Yaralanmalarında Rehabilitasyon. Pelikan Yayıncılık. — https://www.siyasalkitap.com/omuz-yaralanmalarinda-rehabilitasyon
- See also: Başol, O., & Çömlekçi, M. F. (2020). İş tatmini ölçeğinin uyarlanması: Geçerlik ve güvenirlik çalışması. Kırklareli Üniversitesi Sosyal Bilimler Meslek Yüksekokulu Dergisi, 1(2), 17-31. — https://dergipark.org.tr/tr/download/article-file/1442601
- See also: Bat-Erdene, E., Hiramoto, T., Tumurbaatar, E., Tumur-Ochir, G., Jamiyandorj, O., Yamamoto, E., … Lkhagvasuren, B. (2023). Quality of life in the general population of Mongolia: Normative data on WHOQOL-BREF. PLOS ONE, 18(9), e0291427. — https://doi.org/10.1371/journal.pone.0291427
- See also: Baycan, A. (1985). An analysis of several aspects of job satisfaction between different occupational groups. Boğaziçi Üniversitesi. — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=s1KXn1BM2LTQHsVAXojiBw&
- See also: Bhagat, T., Shrestha, A., Acharya, S. K., & Ghimire, U. (2022). Musculoskeletal complaints and associated factors among dental practitioners of Nepal: A nationwide survey. International Journal of Occupational Safety and Ergonomics, 28(4), 2302-2307. — https://pubmed.ncbi.nlm.nih.gov/34615445/
- See also: Bhatia, V., Vaishya, R., Jain, A., Grover, V., Arora, S., Das, G., Saluja, P., & Pandey, H. (2024). Identification of prevalence of musculoskeletal disorders and various risk factors in dentists. Heliyon, 10(1), e24106. — https://pubmed.ncbi.nlm.nih.gov/38332878/
- See also: Chang, L. R., Anand, P., & Varacallo, M. (2025). Anatomy, shoulder and upper limb, glenohumeral joint. In StatPearls. StatPearls Publishing. — https://www.ncbi.nlm.nih.gov/books/NBK537018/
- See also: Cheatham, S. W., Baker, R. T., & Abdenour, T. E. (2021). Kinesiology tape: A descriptive survey of healthcare professionals in the United States. International Journal of Sports Physical Therapy, 16(3), 778-796. — https://pubmed.ncbi.nlm.nih.gov/34123530/
- See also: Çelikel, R., Usgu, G., & Yakut, Y. (2020). The effect of ergonomic education given with physiotherapy program on pain, quality of life and functionality in dentists with wrist pain. Zeugma Journal of Health Researches, 2(2), 82-88. — https://sbf.hku.edu.tr/wp-content/uploads/2020/09/zeugma-health-2-2.pdf
- See also: da Silva, N. C., Chaves, T. C., dos Santos, J. B., Sugano, R. M. M., Barbosa, R. I., Marcolino, A. M., … Fonseca, M. C. R. (2020). Reliability, validity and responsiveness of Brazilian version of QuickDASH. Musculoskeletal Science and Practice, 48, 10216 — https://doi.org/10.1016/j.msksp.2020.102163
- See also: De Sio S, Traversini V, Rinaldo F, et al. Ergonomic risk and preventive measures of musculoskeletal disorders in the dentistry environment: an umbrella review. PeerJ. 2018;6:e4154. doi: 10.7717/peerj.4154 — https://pubmed.ncbi.nlm.nih.gov/29362689/
- See also: Dinibutun, S. R. (2023). Factors affecting burnout and job satisfaction of physicians at public and private hospitals: A comparative analysis. Journal of Healthcare Leadership, 15, 387-401. — https://pubmed.ncbi.nlm.nih.gov/38077693/
- See also: Epperson, T. N., Black, A. C., & Varacallo, M. A. (2023). Anatomy, shoulder and upper limb, sternoclavicular joint. In StatPearls. StatPearls Publishing. — https://www.ncbi.nlm.nih.gov/books/NBK537258/
- See also: Er, G., & Yüksel, İ. (2023). A comparison of the effects of connective tissue massage and classical massage on chronic mechanical low back pain. Medicine, 102(15), e33516. — https://doi.org/10.1097/MD.0000000000033516
- See also: Ergan, M., Ercan, S., İnce Parpucu, T., Başkurt, F., & Başkurt, Z. (2024). Diş hekimliği öğrencilerinin ergonomi ilişkili kas-iskelet sistemi sorunları, kinestezi ve tükenmişlik düzeyleri: Cinsiyete özgü farklılıklar [Ergonomics-related musculoskeletal p — https://doi.org/10.33439/ergonomi.1384047
- See also: Esporlas, B. E., Cervantes, A. P., Banaag, R. T., & De Ramos, B. K. R. P. (2023, November). Hand grip strength of UPHSD College of Dentistry students: A cross-sectional study [Paper presentation]. UPHSD University Week, Las Piñas, Philippines. — https://www.academia.edu/96940283/Handgrip_Force_of_the_Students_of_UPHSD_College_of_Dentistry_A_Sectional_Study?f_ri=966025
- See also: Farha, N. J., Rahmawati, R. S., Ramadhan, G., Manurung, R., Panjaitan, I. T., Olivia, K. L., & Ramadhani, A. (2020). The level of quality of life of preclinic students of dental medicine. Systematic Reviews in Pharmacy, 11(3), 860-863. — https://www.sysrevpharm.org/articles/the-level-of-quality-of-life-of-preclinic-students-of-dental-medicine.pdf
- See also: Faiz, K. W. (2014). VAS-visuell analog skala [VAS-visual analog scale]. Tidsskrift for Den Norske Laegeforening: Tidsskrift for Praktisk Medisin, Ny Raekke, 134(3), 323. — https://doi.org/10.4045/tidsskr.13.1145
- See also: Gandavadi, A., Ramsay, J. R., & Burke, F. J. (2007). Assessment of dental student posture in two seating conditions using RULA methodology-A pilot study. British Dental Journal, *203*(10), 601-605. — https://pubmed.ncbi.nlm.nih.gov/18037853/
- See also: Gibbons, J. (2024). Yaralanma önleme ve yaygın tıbbi durumlar için kinesiyoloji bantlamaya pratik kılavuz (3. baskı). Lotus Publishing. — https://www.scribd.com/document/721897481/A-Practical-Guide-to-Kinesiology-Taping-for-Injury-Prevention-and-Common-Medical-Conditions-John-Gibbons-Z-Library
- See also: Goetti, P., Denard, P. J., Collin, P., Ibrahim, M., Hoffmeyer, P., & Lädermann, A. (2020). Shoulder biomechanics in normal and selected pathological conditions. EFORT Open Reviews, 5(8), 508-518. — https://doi.org/10.1302/2058-5241.5.200006
- See also: Gorce, P., & Jacquier-Bret, J. (2024). Work-related musculoskeletal disorders among surgeons: A bibliometric analysis from 1982 to 2024. Exploration of Musculoskeletal Diseases, 2(4), 317-335. — https://doi.org/10.37349/emd.2024.00059
- See also: Haas, Y., Naser, A., Haenel, J., Fraeulin, L., Holzgreve, F., Erbe, C., … Ohlendorf, D. (2020). Prevalence of self-reported musculoskeletal disorders of the hand and associated conducted therapy approaches among dentists and dental assistants in Germany. — https://doi.org/10.1371/journal.pone.0241564
- See also: Hashim, R., Salah, A., Mayahi, F., & Haidary, S. (2021). Prevalence of postural musculoskeletal symptoms among dental students in United Arab Emirates. BMC Musculoskeletal Disorders, 22(1), 30. — https://doi.org/10.1186/s12891-020-03887-x
- See also: Holzgreve, F., Fraeulin, L., Maurer-Grubinger, C., Betz, W., Erbe, C., Weis, T., ... & Ohlendorf, D. (2022). Effects of resistance training as a behavioural preventive measure on musculoskeletal complaints, maximum strength and ergonomic risk in dentists — https://pubmed.ncbi.nlm.nih.gov/36298418/
- See also: Ilyas, T., Jawa, R., Zulfiqar, H., Maqbool, S., Asghar, H. M. U., & Rehman, A. (2022). Prevalence of upper extremity musculoskeletal problems among male and female dental students: A cross sectional study. Pakistan Journal of Medical & Health Sciences, 1 — https://doi.org/10.53350/pjmhs22167175
- See also: Institute for Work & Health. (2006). QuickDASH - Quick disabilities of the arm, shoulder and hand questionnaire. — https://www.scribd.com/document/498896044/QuickDASH-ftronline
- See also: Kalfoss, M. H., Reidunsdatter, R. J., Klöckner, C. A., & Nilsen, M. (2021). Validation of the WHOQOL-Bref: Psychometric properties and normative data for the Norwegian general population. Health and Quality of Life Outcomes, 19(1), 13. — https://doi.org/10.1186/s12955-020-01656-x
- See also: Kawtharani, A. A., Chemeisani, A., Salman, F., Haj Younes, A., & Msheik, A. (2023). Neck and musculoskeletal pain among dentists: A review of the literature. Cureus, 15(1), e33609. — https://doi.org/10.7759/cureus.33609
- See also: Kerosuo, E., Kerosuo, H., & Kanerva, L. (2000). Self-reported health complaints among general dental practitioners, orthodontists, and office employees. Acta Odontologica Scandinavica, 58(5), 207-212. — https://doi.org/10.1080/000163500750051755
- See also: Koldas Dogan S, Ay S, Evcik D, Baser O. Adaptation of Turkish version of the questionnaire Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) in patients with carpal tunnel syndrome. Clin Rheumatol. 2011 Feb;30(2):185-91. doi: 10.1007/s10067-01 — https://pubmed.ncbi.nlm.nih.gov/20411289/
- See also: Kumbrink, B. (2014). Spesifik endikasyonlar için uygulamalar, impingement sendromu. G. Yapalı (Ed.), K-taping içinde (s. 135). Hipokrat Kitabevi. — https://link.springer.com/chapter/10.1007/978-3-662-43573-1_1
- See also: Labriola, J. E., Lee, T. Q., Debski, R. E., & McMahon, P. J. (2005). Glenohumeral eklemin stabilitesi ve instabilitesi: omuz kaslarının rolü [Stability and instability of the glenohumeral joint: The role of shoulder muscles]. Journal of Shoulder and Elbo — https://doi.org/10.1016/j.jse.2004.09.014
- See also: Maier, S. P., II, Rudisill, S. S., Wright, C. L., Daniell, H. D., Lydston, M., & O'Donnell, E. A. (2022). Sex differences in shoulder anatomy and biomechanics: A systematic review and meta-analysis. Journal of Women's Sports Medicine, 2(1), 5-17. — https://doi.org/10.53646/jwsm.v2i1.19
- See also: McCausland, C., Sawyer, E., Eovaldi, B. J., & Varacallo, M. (2023). Anatomy, shoulder and upper limb, shoulder muscles. In StatPearls. StatPearls Publishing. — https://www.ncbi.nlm.nih.gov/books/NBK534836/
- See also: Moodley R, Naidoo S, Wyk JV. The prevalence of occupational health-related problems in dentistry: a review of the literature. J Occup Health. 2018;60(2):111-125. doi: 10.1539/joh.17-0188-RA — https://pubmed.ncbi.nlm.nih.gov/29213011/
- See also: Nalbantoğlu, C. B. (2012). Yükseköğretim kurumlarında akademisyenlerin örgütsel bağlılığının iş tatminine etkisi: Plato Meslek Yüksekokulu, Beykoz Lojistik Meslek Yüksekokulu, Beykent Üniversitesi saha araştırması [Yüksek lisans tezi]. İstanbul Aydın Ü — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=9LhlOV_Rtx06SuuMLZ9NUA&no=Ocy-bMJCWNvvAm9iMJT5fg
- See also: Partovi, A. (2020). Assessment of awareness and attitude of dental ergonomics among international students [Unpublished master's thesis]. Lithuanian University of Health Sciences. — https://portalcris.lsmuni.lt/server/api/core/bitstreams/b37cbe5e-8259-407f-a45c-14b0f3e8d7d3/content
- See also: Pejčić, N., Petrović, V., Đurić-Jovičić, M., Medojević, N., & Nikodijević-Latinović, A. (2021). Analysis and prevention of ergonomic risk factors among dental students. European Journal of Dental Education, 25(3), 460-479. — https://doi.org/10.1111/eje.12621
- See also: Perry, C. M., & Lippincott, E. L. (2020). The effects of kinesiology tape on shoulder stability and functional performance. Keystone Undergraduate Research Journal, 7(1), 1-6. — https://www.ship.edu/globalassets/keystone-journal/v7n1_perry_lippincott.pdf
- See also: Porcellini, G., Caranzano, F., Campi, F., Pellegrini, A., & Paladini, P. (2011). Glenohumeral instabilite ve rotator manşet yırtığı [Glenohumeral instability and rotator cuff tear]. Sports Medicine and Arthroscopy Review, 19, 395-400. — https://pubmed.ncbi.nlm.nih.gov/22089289/
- See also: Ray, B., Patil, S., & Savant, A. (2021). Effect of cognitive ability on oral health status: A scoping review of observational studies. Journal of Oral Biology and Craniofacial Research, 11(4), 574-579. — https://doi.org/10.1016/j.jobcr.2021.07.007
- See also: Rickert, C., Fels, U., Gosheger, G., Kalisch, T., Liem, D., Klingebiel, S., Schneider, K. N., & Schorn, D. (2021). Prevalence of musculoskeletal diseases of the upper extremity among dental professionals in Germany. Risk Management and Healthcare Policy, — https://doi.org/10.2147/RMHP.S316795
- See also: Shah, M., & Patil, C. (2024). Additive effect of kinesiotaping on neck pain and grip strength in violin players: An experimental study. International Journal of Health Sciences and Research, 14(4), 129-139. — https://doi.org/10.52403/ijhsr.20240419
- See also: Soylu, M., & Altındiş, S. (2018). Diş hekimlerinin çalışma şartlarının mesleki kas-iskelet sistemi hastalıklarına etkisi [The effect of working conditions of dentists on occupational musculoskeletal system diseases]. SDÜ Sağlık Bilimleri Enstitüsü Dergis — https://dergipark.org.tr/tr/download/article-file/458799
- See also: Suzuk, E. (2020). Sağlık çalışanlarının inanç düzeylerinin iş doyumuna etkisi [Yayımlanmış yüksek lisans tezi]. Selçuk Üniversitesi. — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=a1vkixubgo88UNEMab6x9g&no=6qMoAdc4RM6syh2fXrLnQA
- See also: Türkiye Psikiyatri Derneği. (t.y.). WHOQOL-BREF (TR). 20 Aralık 2024 tarihinde — https://psikiyatri.org.tr/uploadFiles/whoqolbrief.pdf
- See also: Valachi, B., & Valachi, K. (2003). Preventing musculoskeletal disorders in clinical dentistry: Strategies to address the mechanisms leading to musculoskeletal disorders. Journal of the American Dental Association, 134(12), 1604-1612. — https://pubmed.ncbi.nlm.nih.gov/14719757/